CLINICAL TRIAL: NCT00104247
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Phenoptin™ in Subjects With Phenylketonuria Who Have Elevated Phenylalanine Levels
Brief Title: Study to Evaluate the Safety and Efficacy of Phenoptin™ in Subjects With Phenylketonuria Who Have Elevated Phenylalanine Levels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKU-003
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Results first posted 2009-04-16 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Phenylketonurias
Keywords: Phenylalanine Hydroxylase
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

INTERVENTIONS:
Drug: sapropterin dihydrochloride, 6R-BH4, tetrahydrobiopterin

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Phenoptin™ (sapropterin dihydrochloride) in reducing blood phenylalanine (Phe) levels in subjects with phenylketonuria.

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age and older
* Received at least 7 out of 8 scheduled doses in Study PKU 001
* Responsive to Phenoptin™ in Study PKU-001, defined as a reduction in blood Phenylalanine level of >/=30% compared with baseline
* Blood Phenylalanine level >/=450 μmol/L at screening
* Willing and able to provide written informed consent or, in the case of subjects under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained
* Negative urine pregnancy test at screening (females of child-bearing potential)
* Male and Female subjects of childbearing potential (if sexually active) must be using acceptable birth control measures, as determined by the investigator, and willing to continue to use acceptable birth control measures while participating in the study
* Willing and able to comply with study procedures
* Willing to continue current diet unchanged while participating in the study

Exclusion Criteria:

* Perceived to be unreliable or unavailable for study participation or, if under the age of 18, have parents or legal guardians who are perceived to be unreliable or unavailable
* Use of any investigational agent other than Phenoptin™ within 30 days prior to screening, or requirement for any investigational agent or investigational vaccine prior to completion of all scheduled study assessments
* Pregnant or breastfeeding, or considering pregnancy
* ALT >5 times the upper limit of normal (i.e., Grade 3 or higher based on World Health Organization Toxicity Criteria) at screening
* Concurrent disease or condition that would interfere with study participation or safety (e.g., seizure disorder, oral steroid-dependent asthma or other condition requiring oral or parenteral corticosteroid administration, or insulin-dependent diabetes, or organ transplantation recipient)
* Serious neuropsychiatric illness (e.g., major depression) not currently under medical management
* Requirement for concomitant treatment with any drug known to inhibit folate synthesis (e.g., methotrexate)
* Concurrent use of levodopa
* Clinical diagnosis of primary BH4 deficiency

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-03; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Los Angeles, California
  - Oakland, California
  - New Haven, Connecticut
  - Chicago, Illinois
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin

REFERENCES:
- [Derived] Levy HL, Milanowski A, Chakrapani A, Cleary M, Lee P, Trefz FK, Whitley CB, Feillet F, Feigenbaum AS, Bebchuk JD, Christ-Schmidt H, Dorenbaum A; Sapropterin Research Group. Efficacy of sapropterin dihydrochloride (tetrahydrobiopterin, 6R-BH4) for reduction of phenylalanine concentration in patients with phenylketonuria: a phase III randomised placebo-controlled study. Lancet. 2007 Aug 11;370(9586):504-10. doi: 10.1016/S0140-6736(07)61234-3. PMID 17693179
- See also: BioMarin Pharmaceutical Inc. home page — http://www.bmrn.com
- See also: NDA Review Package — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails
- See also: Product Label — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Label_ApprovalHistory

RESULTS

PARTICIPANT FLOW:
Groups:
- Sapropterin Dihydrochloride: Patients administered 10 mg /kg orally once daily.
- Placebo: Placebo
Period: Overall Study
Arm/Group | Sapropterin Dihydrochloride | Placebo
Started | 42 | 47
Completed | 41 (Subject withdrew prior to dosing) | 46 (One subject withdrew at Week 4, but is included in the data analysis)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Noncompliant with dosing | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sapropterin Dihydrochloride | Placebo | Total
Number analyzed (Participants) | 41 | 47 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (9.5) | 19.5 (9.8) | 20.4 (9.7)
Age, Customized [Number; unit: Years]
  8 <= Age <= 12 | 6 | 11 | 17
  12 < Age | 35 | 36 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 37
  Male | 27 | 24 | 51
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Pacific Islander | 1 | 0 | 1
  Caucasian | 39 | 47 | 86
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Phenylalanine Levels From Baseline to Week 6.
Time Frame: baseline to week 6
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Sapropterin Dihydrochloride | Placebo
Number analyzed (Participants) | 41 | 46
micromole per liter
  Baseline Blood Phe Level | 843 (300) | 888 (323)
  Week 6 Blood Phe Level | 607 (377) | 891 (348)
  Mean Change in Blood Phe from Baseline to Week 6 | -239 (38) | 6 (36)
Statistical Analysis 1: Comparison: Sapropterin Dihydrochloride vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Arm/Group | Sapropterin Dihydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/47
Other Adverse Events (participants affected / at risk) | 21 | 34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sapropterin Dihydrochloride | Placebo
Upper Respiratory Tract Infection (Infections and infestations) | 7/41 | 13/47
Pharyngitis (Infections and infestations) | 2/41 | 1/47
Infection (Infections and infestations) | 2/41 | 0/47
Vomiting (Gastrointestinal disorders) | 2/41 | 4/47
Abdominal Pain (Gastrointestinal disorders) | 1/41 | 4/47
Diarrhoea (Gastrointestinal disorders) | 2/41 | 3/47
Headache (Nervous system disorders) | 4/41 | 7/47
Pyrexia (General disorders) | 2/41 | 2/47
Back Pain (Musculoskeletal and connective tissue disorders) | 1/41 | 3/47
Cough (Respiratory, thoracic and mediastinal disorders) | 0/41 | 3/47
Pharynholaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3/41 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results shall be made by Sponsor in a joint publication. If such a multi-center publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from their site individually, subject however to comply with the other terms of the agreement.